CLINICAL TRIAL: NCT07081334
Title: Phase 1 Study to Assess the Safety and Exploratory Immunogenicity of PV-001
Brief Title: A Phase 1 Study of PV-001 9-valent Human Papillomavirus(HPV) Vaccine
Acronym: HPV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POSVAX (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: POCLI-101
Record Dates: First submitted 2025-06-30; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: HPV Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PV-001 vaccine (Experimental)
  Interventions: Biological: PV-001
- PEV-001 (Placebo Comparator)
  Interventions: Biological: PEV-001

INTERVENTIONS:
Biological: PV-001 — 9-valent vaccine containing antigens for HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58
  Arms: PV-001 vaccine
Biological: PEV-001 — PEV-001 is a formulation of the PV-001 vaccine that excludes the HPV antigens and contains only aluminum phosphate.
  Arms: PEV-001

SUMMARY:
Study Title:

Evaluation of the Safety and Immunogenicity of a Third Dose of PV-001 in Healthy Women Aged 19-45

Objective:

To assess the safety and antibody response of a third dose of PV-001 in healthy adult female participants.

Key Questions Is PV-001 safe? What adverse events may occur after vaccination? Does PV-001 produce an effective immune response?

Participant Activities :

Three clinic visits for screening and vaccination Blood samples collected on a set schedule Monitoring for side effects after vaccination

ELIGIBILITY:
1. Inclusion criteria

   * Healthy women between the ages of 19 and 45 years old
   * Able to comply with the planned visit schedule for this study to perform the study procedures
   * Able to understand and complete the immunization diary provided in this study
   * Able to have a specimen collected and tested for a Pap test
   * Have been using contraception for 48 hours prior to the screening visit and are able to maintain contraception for the duration of the study
   * After receiving and understanding a detailed explanation of this study, they have voluntarily decided to participate and have given written informed consent.
2. Exclusion criteria

   * Previous HPV vaccination or participation in a clinical trial of HPV vaccine
   * Previous history of abnormal pap test or colposcopy with abnormal cervical cells
   * Previous HPV test positive for one or more of the following types: HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58, or positive human papillomavirus genotyping test at screening
   * Acute fever (38.0°C or higher) within 24 hours prior to the first dose of the investigational medicinal product
   * Positive results of viral tests [hepatitis B test, human immunodeficiency virus (HIV) test, hepatitis C test] at screening or suspected of infection
   * Subjects with clinically significant abnormal results of clinical laboratory tests at screening, as judged by the investigator
   * Immune response is impaired by genetic defects, human immunodeficiency virus (HIV) infection, or other causes.
   * Have a history of neurological disease, such as encephalomyelitis or Guillain-Barre syndrome
   * History of HPV-related malignancy (cervical cancer, vulvar cancer, vaginal cancer, anal cancer, genital warts, cervical intraepithelial adenocarcinoma, cervical intraepithelial neoplasia, vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, anal intraepithelial neoplasia)
   * Received Immunosuppressive Therapy including radiotherapy, antimetabolites, alkylating agents, cytotoxic agents, or cytotoxic agents within 1 year prior to the first dose of investigational medicinal product.
   * Have received an immunosuppressant or immune modifying drug within 6 months prior to the first dose of the investigational drug.

     1. Azathioprine, Cyclosporin, Interferon, G-CSF, Tacrolimus, Everolimus, Sirolimus, etc.
     2. High doses of systemic steroids: Corticosteroids up to 2 mg/kg/day based on Prednisolone or doses of 20 mg/day or more used continuously for more than 14 days are considered high doses and excluded from participation in this study. However, Inhaled, Nasal, Conjunctiva, Intraarticular, Bursal, or Tendon injections, and Topical corticosteroids are allowed regardless of dose.
     3. Administration of immunoglobulins or blood-derived products within 3 months prior to the first dose of investigational medication
     4. Have thrombocytopenia, blood coagulation disorders at risk of causing serious bleeding or have received anticoagulants* within 3 weeks prior to Visit 2

        * Anticoagulants: anticoagulants such as coumarin/warfarin or new oral anticoagulants/antiplatelet agents
     5. Have or have had a history of myocardial infarction
     6. Have had anaphylaxis or serious adverse events related to the vaccine
     7. Hypersensitivity to any investigational drug or component (including aluminum, yeast)
     8. History of alcohol or other substance abuse
     9. History of malignancy
     10. Have a serious acute, chronic, or progressive medical condition (e.g., malignancy, cardiovascular, respiratory, endocrine, renal, or hepatic disease, etc.) that, in the opinion of the investigator, may interfere with the progress and completion of this study
     11. History of vaccination with any other vaccine within 4 weeks prior to the first dose of the investigational drug or planned vaccination with any other vaccine within 4 weeks after each dose of the investigational drug.
     12. Women of childbearing potential who do not agree to use a medically acceptable method of contraception for the duration of the study (hormonal contraception, intrauterine device (IUD) or intrauterine system (IUS), tubal ligation, double barrier method (combined use such as cervical cap, contraceptive diaphragm with male condom)
     13. Pregnant or lactating women
     14. Subjects who have received another investigational drug within 6 months prior to the first dose of the investigational drug or who are scheduled to receive another investigational drug during the study
     15. For any other reason, the investigator considers you unsuitable to be a subject in this study.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Safety assessment | 180 days after last dose of vaccination
  Adverse Events:
  Immediate adverse reactions occurring within 30 minutes after administration of the investigational product (e.g., syncope, loss of consciousness, anaphylaxis-related events),
  Expected local and systemic adverse reactions occurring within 7 days following administration of the investigational product, and
  Unexpected adverse events occurring from the first dose through 180 days after the third dose (Visit 11).

SECONDARY OUTCOMES:
Exploratory immunogenicity assessment | At 4 months after the second dose (Visit 8) and 28 days after the third dose (Visit 10), relative to baseline (Visit 1, prior to the first dose of the investigational product)
  Antibody titers (GMTs) and fold increases (GMRs), measured by ELISA, will be evaluated at 4 months after the second dose and 28 days after the third dose, relative to baseline levels assessed prior to the first dose of the investigational product.
  Neutralizing antibody titers (GMTs) and fold increases (GMRs) against HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 will be measured using a pseudovirus-based neutralization assay at 4 months after the second dose (Visit 8) and 28 days after the third dose (Visit 10), relative to baseline levels measured prior to the first dose of the investigational product (Visit 1).

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim JH, Lee YK, Cho HB, Choi JW, Mun GI, Song OG, Hong J, Kim HJ, Lee A, Choo S, Kim HJ. Evaluation of the safety and immunogenicity of a 9-valent human papillomavirus vaccine produced in Saccharomyces cerevisiae using a heating-chilling process for virus-like particle antigen assembly: a double-blind, randomized, placebo-controlled phase 1 clinical trial. Lancet Reg Health West Pac. 2025 Sep 19;62:101686. doi: 10.1016/j.lanwpc.2025.101686. eCollection 2025 Sep. PMID 41048471